CLINICAL TRIAL: NCT06148766
Title: An Investigation of the Effects of a Royal Jelly and Bee Venom-Derived Skin Cream on Skin Health and Signs of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuka Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20378
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Skin Health
MeSH Terms: interventions — royal jelly; Bee Venoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eternal Renewal Regenerating Face Cream (Experimental): Participants will be required to apply the test product in the morning and before bedtime at night.
  After thoroughly cleansing and toning the face, the participants will take a pea-sized amount of face cream and apply it to the face, massaging over the entire face with small circular movements until the cream has fully absorbed.
  Interventions: Other: Manuka Health Eternal Renewal Regenerating Face Cream with Royal Jelly and Bee Venom

INTERVENTIONS:
Other: Manuka Health Eternal Renewal Regenerating Face Cream with Royal Jelly and Bee Venom — Face cream containing manuka honey, royal bee jelly, and bee venom.

SUMMARY:
This is a virtual, single-group clinical trial that will last 8 weeks. Participants will use the Manuka Health Eternal Renewal Regenerating Face Cream with Royal Jelly and Bee Venom twice daily and complete questionnaires at Baseline, Week 2, Week 4, and Week 8.

Participants will also undergo skin analysis via the Optic Elite facial skin analysis system at Baseline and Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* 40-55 years of age.
* Must be in good general health.
* Must have concerns with overall skin health and appearance, including:

Fine lines and wrinkles The appearance of dark spots

* Must be using the same cleanser and toner for at least one month prior to starting the study.
* Must be willing to keep using the same cleanser and toner for the duration of the study.
* Must not be using oral or topical retinoids.
* In the last three months, has not introduced any new medications or supplements that target skin health.
* Must be willing to comply with the protocol.

Exclusion Criteria:

* Anyone with an allergy to bees or bee products.
* Females who are pregnant or breastfeeding.
* Unwilling to follow the protocol.
* Unwilling to maintain use of the same cleaner and toner for the duration of the study.
* Currently participating in another study.
* Use of oral or topical retinoids.
* Individuals with cystic acne or otherwise self-reported very acne-prone skin.
* Use of a prescription medication relevant to the skin.
* Anyone undergoing cosmetic procedures during the study, including Botox, laser, or chemical peel treatments.
* Anyone sensitive or allergic to any ingredients found in the products.
* Anyone with severe chronic conditions, including oncological conditions, psychiatric disorders or diabetes.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in signs of skin health over time assessed via Optic Elite Skin Analysis. [Timeframe: Baseline to Week 8] | 8 weeks
  The Optic Elite skin analysis system clinically measures the surface and subsurface layers of skin using digital imaging technology

SECONDARY OUTCOMES:
Changes in self-perceived appearance of fine lines and wrinkles. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin clarity. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin hydration. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin texture. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin hyperpigmentation. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin irritation. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin brightness. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin tone evenness. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided